CLINICAL TRIAL: NCT04828694
Title: A Randomized, Open Label, Single Dose Pharmacokinetic and Safety Study of Implantable Long Acting 3-month Naltrexone Subcutaneous Pellets Compared to Naltrexone IM Injection (Vivitrol) in Healthy Volunteers
Brief Title: Pharmacokinetic and Safety Study of Naltrexone Release From Subcutaneous BICX104 Pellets Compared to Vivitrol Injections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCorRx Inc (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The HEAL Initiative (https://heal.nih.gov/) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BioCorRx-21-01a; UG3DA047925 (NIH)
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BICX104 (Experimental): BICX104 is an eroding implantable pellet that contains 1 g naltrexone and 11 mg magnesium stearate that will be inserted subcutaneously. It will be administered once for 84 days.
  Interventions: Drug: BICX104
- Vivitrol (Active Comparator): Vivitrol intramuscular injection containing 380 mg of naltrexone. Three consecutive doses will be administered once every 28 days for 84 days.
  Interventions: Drug: Vivitrol

INTERVENTIONS:
Drug: BICX104 — Erodable implantable pellet containing 1 g naltrexone and 11 mg magnesium stearate.
  Arms: BICX104
Drug: Vivitrol — Intramuscular injection containing 380 mg of naltrexone.
  Arms: Vivitrol

SUMMARY:
This is a Phase 1, 6-month, open-label, multi-center study in parallel groups of randomized healthy volunteers to evaluate the pharmacokinetics and safety of BICX104 implantable subcutaneous naltrexone pellets and Vivitrol intramuscular depot naltrexone injection.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Female or male subjects aged 18-50 years old.
3. Without current non-remitted DSM-5 (The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) - Substance Use Disorders diagnoses; subjects with a sustained remission diagnosis are not excluded.
4. In good health, as determined by the study physician, based on complete medical history, physical examination, vital signs measurement, ECG, and laboratory tests within normal ranges, to permit treatment.
5. Weight of 100-180 pounds, and a BMI of 18.5 to 30 kg/m2, inclusive.
6. Must agree to comply with all study requirements and be willing to complete entire study.
7. Females of childbearing potential and males willing to practice an effective method(s) of birth control for the duration of participation in the study (<1% failure rate per year).

Exclusion Criteria:

1. Is pregnant, is planning to become pregnant or breastfeed infants during the study.
2. Is currently treated with naltrexone or has had a naltrexone implant in the past 2 years or received Vivitrol treatment in the past year.
3. Clinically significant medical/psychological condition or abnormality at screening (i.e., physical examination, electrocardiogram [ECG], hematology or blood chemistry evaluation, or urinalysis findings), including any diagnosis of Hepatitis B, Hepatitis C or HIV infection.
4. Presence of opiates, cocaine, methamphetamine or other significant drugs of abuse in the urine (as determined by urine drug test).
5. Any active hepatitis or hepatic failure or dysfunction evidenced by the following: aspartate transaminase (AST) or alanine transaminase (ALT) higher than 1.5 times the upper limit of normal (1.5xULN), hyperbilirubinemia (bilirubin >10% above ULN), creatine phosphokinase (CPK) higher than 2.5xULN, prolonged prothrombin time (international normalized ratio ≥1.7), ascites, or esophageal variceal disease.
6. Manifestation of suicidal ideation, psychotic symptoms (including significant violent behavior), or psychiatric or neurological disorders that would compromise ability to complete the study.
7. Participation in a methadone program currently or within past 3 years, or 3 or more previous medically supervised detoxification treatments in past 3 years.
8. If a healthy volunteer fails one naloxone challenge, the subject will not be suitable for the study. The only exceptions will be made when a 'false positive' test result is received for the first test.
9. Intolerance and/or hypersensitivity to naltrexone, naloxone, or polylactide-co-polymers such as polylactide-co-glycolide (PLG).
10. Participation in a clinical trial within 30 days of screening.
11. Has a condition which requires or may require treatment with opioid based medication.
12. Is prone to skin rashes, irritation or has a chronic skin condition.
13. Alcohol Use Disorder diagnosis.
14. Has a predisposition to poor response to an implant site reaction, as judged by the study physician.
15. Has a history of keloid formation, connective tissue disease, e.g., scleroderma, or history of recurrent MRSA infections.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Cmax. | 140 Days
  Maximum observed mean plasma concentration [Cmax] of naltrexone and 6-beta-naltrexol.
Pharmacokinetic parameter: Tmax. | 140 Days
  Time to mean maximum observed drug concentration (Tmax) of naltrexone and 6-beta-naltrexol.
Pharmacokinetic parameter: Css. | 140 Days
  Changes in the mean observed steady state plasma concentration [Css] of naltrexone and 6-beta-naltrexol.
Pharmacokinetic parameter: AUC | 140 Days
  Area Under the Plasma Concentration Versus Time Curve (AUC) of naltrexone and 6-beta-naltrexol.
Pharmacokinetic parameter: Tlast ≥ 1ng/ml naltrexone. | 140 Days
  Time of Last Quantifiable Plasma Concentration (Tlast) of naltrexone greater than or equal to 1ng/ml.
Pharmacokinetic parameter: Tlast. | 140 Days
  Time of Last Quantifiable Plasma Concentration (Tlast) of naltrexone and 6-beta-naltrexol.

SECONDARY OUTCOMES:
Safety Parameter: AEs | 168 Days
  Incidence and severity of adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No